CLINICAL TRIAL: NCT05724134
Title: Role of Hyperinsulinemia in Non-Alcoholic Fatty Liver Disease (NAFLD) Pathogenesis: Pancreatic Clamp Pilot & Feasibility Study
Brief Title: Pancreatic Clamp in NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Albert Einstein College of Medicine (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAU3014; 3P30DK063608 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance; Prediabetic State; Hyperinsulinemia; Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: Insulin resistance; Hyperinsulinemia; Diabetes; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Insulin Resistance; Prediabetic State; Hyperinsulinism; Non-alcoholic Fatty Liver Disease; Obesity; Diabetes Mellitus | interventions — Insulin; Octreotide; Glucagon; Human Growth Hormone; Glucose

STUDY DESIGN:
Intervention Model Description: All participants will undergo (i.e., cross over between) both pancreatic clamp protocols (MH, RE) separated by 2-8 weeks. The order of the clamp protocols (i.e., MH > RE, RE > MH) will be randomized.
Who Masked: Participant
Masking Description: Participant will be blinded to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Maintenance hyperinsulinemia (MH) protocol (Active Comparator): The basal insulin infusion rate (IIR) necessary to maintain participants' mean basal fasting plasma glucose (mbFPG) will be determined during the basal titration period. Then, during the intervention period, the IIR will remain at 100% of basal for the full duration (225 min). The IIR and resulting insulin levels are expected to be relatively high (cf. hyperinsulinemia) because of underlying insulin resistance.
  Interventions: Drug: Insulin human; Drug: Octreotide Acetate; Drug: Glucagon; Drug: Growth Hormone, Human; Other: [6,6-2H2] D-glucose; Drug: 20% D-glucose (aq); Dietary Supplement: BOOST Plus; Dietary Supplement: CORE Bar; Device: Harvard Apparatus PHD ULTRA CP syringe pump; Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer
- Reduction toward euinsulinemia (RE) protocol (Experimental): The basal insulin infusion rate (IIR) necessary to maintain participants' mean basal fasting plasma glucose (mbFPG) will be determined during the basal titration period. Then, during the intervention period, the basal IIR will be reduced by up to 50%. Thus, the basal hyperinsulinemia expected due to underlying insulin resistance will be reduced toward euinsulinemia.
  Interventions: Drug: Insulin human; Drug: Octreotide Acetate; Drug: Glucagon; Drug: Growth Hormone, Human; Other: [6,6-2H2] D-glucose; Drug: 20% D-glucose (aq); Dietary Supplement: BOOST Plus; Dietary Supplement: CORE Bar; Device: Harvard Apparatus PHD ULTRA CP syringe pump; Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer

INTERVENTIONS:
Drug: Insulin human — Insulin infusion rate (IIR) will be determined empirically first to maintain mean basal fasting plasma glucose, and then either maintained at the basal rate (MH protocol) or be reduced stepwise toward euinsulinemia (RE protocol).
Drug: Octreotide Acetate — Octreotide will be infused at 30 ng/kg/min to suppress endogenous insulin, glucagon, and growth hormone secretion. Co-administered with glucagon and rhGH.
Drug: Glucagon — Glucagon will be replaced at a constant rate of up to 0.65 ng/kg/min to maintain baseline counterregulatory response. Co-administered with octreotide and rhGH.
Drug: Growth Hormone, Human — Recombinant human growth hormone (rhGH) will be replaced at a constant rate of up to 3 ng/kg/min to maintain baseline counterregulatory response. Co-administered with octreotide and glucagon.
Other: [6,6-2H2] D-glucose — Stable isotope tracer administered to calculate glucose kinetics during pancreatic clamp.
  Other Names: D2-glucose, D2G
Drug: 20% D-glucose (aq) — 20% D-glucose (aq) (D20W) will be administered to counteract hypoglycemia or strongly downward blood glucose trends, as needed.
  Other Names: D20W
Dietary Supplement: BOOST Plus — Nutritional supplement will be administered to provide three standardized "mixed meals" on the day before the pancreatic clamp.
Dietary Supplement: CORE Bar — Energy bar used as a standardized snack on the day before the pancreatic clamp.
Device: Harvard Apparatus PHD ULTRA CP syringe pump — Syringe pump used for highly precise administration of insulin, octreotide/glucagon/rhGH, and D20W (as needed) even at low infusion rates.
Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer — Glucose oxidase analyzer used to detect plasma glucose levels at the point of care. YSI have been the gold standard in clamp studies for many years. Two machines will run in parallel to ensure accuracy of results.

SUMMARY:
This is a single-center, prospective, randomized, controlled (crossover) clinical study designed to investigate the specific dose-response impact of insulin infusion rate (IIR) on blood glucose levels during a pancreatic clamp study. The investigators will recruit participants with a history of overweight/obesity and evidence of insulin resistance (i.e., fasting hyperinsulinemia plus prediabetes and/or impaired fasting glucose and/or Homeostasis Model Assessment of Insulin Resistance [HOMA-IR] score >=2.73), and with evidence of, or clinically judged to be at high risk for, uncomplicated non-alcoholic fatty liver disease (NAFLD). Participants will undergo two pancreatic clamp procedures in which individualized basal IIR are identified, followed in one by maintenance of basal IIR (maintenance hyperinsulinemia, MH) and in the other by a stepped decline in IIR (reduction toward euinsulinemia, RE). In both clamps the investigators will closely monitor plasma glucose and various metabolic parameters. The primary outcome will be the absolute and relative changes in steady-state plasma glucose levels at each stepped decline in IIR.

DETAILED DESCRIPTION:
Although high blood sugar and risk of heart disease are the most well-known health effects of type 2 diabetes (T2DM), nonalcoholic fatty liver disease (NAFLD), in which too much fat accumulates in the liver, has come to be recognized as another important complication. Unchecked, NAFLD can progress to severe liver inflammation, liver failure, and even liver cancer. The investigators suspect that high levels of the blood sugar-lowering hormone insulin leads to excessive fat production by the liver, and so lowering insulin levels might help to improve NAFLD. In order to answer this question, the investigators will recruit people at risk for T2DM and NAFLD to perform a "pancreatic clamp" - a procedure in which the body's production of insulin is temporarily shut off and then replaced at the same or lower levels. Again, the investigators expect that lowering insulin levels will lower fat production. Because this is a new research approach, the investigators first need to understand how lowering insulin levels affects blood sugar. Research participants in this pilot study will therefore undergo two pancreatic clamps in random order: one roughly maintaining their own internal ("basal") insulin level and one in which the investigators lower that basal insulin level by up to 50%. In each case, the investigators will observe the absolute and relative changes in blood sugar and the levels of certain fats as the investigators change the insulin level. Once the investigators have found a lower insulin level that they can safely maintain, the investigators will go on to study its effect on fat production in a later study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (using highly effective contraception if of childbearing potential, aged 18-65 years
2. Body mass index of 25-45 kg/m2
3. Able to understand written and spoken English and/or Spanish
4. Evidence of insulin resistance, represented by any or all of the following criteria:

   a. Meeting either of the American Diabetes Association's definitions for prediabetes or IFG within the previous year* and on screening labs: i. Prediabetes: Hemoglobin A1c 5.7-6.4% ii. IFG: plasma glucose of 100-125 mg dL-1 after 8-h fast b. Homeostasis Model of Insulin Resistance (HOMA-IR) score ≥ 2.73
5. Fasting hyperinsulinemia (fasting insulin level ≥ 13 µIU/mL) on screening labs
6. Diagnosed with, or clinically judged to be at high risk for, non-alcoholic fatty liver disease (NAFLD), also known as metabolic-associated fatty liver disease (MAFLD), by hepatologist or other qualified specialist physician and the condition is listed as an active problem in the electronic medical record
7. Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Unable to provide informed consent in English or Spanish
2. Concerns arising at screening visit (any of the following):

   i. Unwillingness to use only bedpan or urinal to void during the clamp

   ii. Unwillingness to fast (except water) for up to 22 hours

   iii. Documented weight loss of ≥ 5% of baseline within the previous 6 months

   iv. Abnormal blood pressure (including on treatment, if prescribed)
   * Systolic blood pressure < 90 mm Hg or > 160 mm Hg, and/or
   * Diastolic blood pressure < 60 mm Hg or > 100 mm Hg

     v. Abnormal resting heart rate: <60 or ≥100 bpm
   * Sinus brady- or tachycardia that has been extensively worked up and considered benign by the recruit's personal physician may be permitted at the Principal Investigator's discretion

   vi. Abnormal screening electrocardiogram (or if on file, performed within previous 90 d)
   * Non-sinus rhythm
   * Significant corrected QT segment (QTc) prolongation (≥ 480 ms)
   * New or previously unknown ischemic changes that persist on repeat EKG: 1. ST segment elevations; 2. T-wave inversions

   vii. Laboratory evidence of diabetes mellitus:
   * Hemoglobin A1c ≥ 6.5%, and/or
   * Fasting plasma glucose ≥ 126 mg/dL

   viii. Positive qualitative β-hCG (i.e., pregnancy test) in women of childbearing potential

   ix. Liver function abnormalities (either of the following) - Transaminases (AST or ALT) > 3.0 x the upper limit of normal - Total bilirubin > 1.25 x the upper limit of normal

   x. Abnormal fasting triglycerides at screening ≥ 400 mg/dL

   xi. Abnormal screening serum electrolytes (any of the following)
   * Sodium, potassium, or bicarbonate outside of the reference range
   * Creatinine equating to estimated glomerular filtration rate < 60 mL min-1 1.73 m-2

   xii. Abnormal complete blood count (CBC) (any of the following)
   * Hemoglobin < 10 g dL-1 or hematocrit < 30%
   * Platelet count < 100,000 µL-1
   * Exempt from CBC requirement if previously obtained value within 2 months of screening is available
3. Unwillingness to comply with masking and COVID-19 testing requirements per NYP/CUMC policy
4. Reproductive concerns i. Women of childbearing potential not using highly effective contraception, defined as:

   * Surgical sterilization (e.g., bilateral tubal occlusion, bilateral oophorectomy and/or salpingectomy, hysterectomy)
   * Combined oral contraceptive pills taken daily, including during the study
   * Intrauterine device (levonorgestrel-eluting or copper) active at the time of study
   * Medroxyprogesterone acetate (Depo-Provera®) injection active at the time of study
   * Etonogestrel implants (e.g., Implanon®, etc.) active at the time of the study
   * Norelgestromin/ethinyl estradiol transdermal system (e.g., Ortho-Evra®) active at the time of the study

   ii. Women currently pregnant, measured by serum and/or urine human chorionic gonadotropin, beta subunit (β-hCG)

   iii. Women currently breastfeeding
5. Concerns related to glucose metabolism i. History of having met any of the American Diabetes Association's definitions of diabetes mellitus (i.e., overt diabetes) ii. History of gestational diabetes mellitus within the previous 5 years iii. Use of antidiabetic medications other than metformin within the 90 days prior to screening, including those prescribed for other indications (e.g., weight control, restoration of ovulation in of polycystic ovarian syndrome) iv. Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease) v. Fasting plasma glucose < 89 mg/dL at screening
6. Concerns related to lipid metabolism i. Known diagnoses of familial hypercholesterolemia, familial combined hyperlipidemia, or familial hyperchylomicronemia in the participant or a first-degree relative ii. Use of certain lipid-lowering drugs other than statins for primary prevention within 90 d prior to screening visit, including: • Statins or PCSK9 inhibitors for secondary prevention or treatment of familial hypercholesterolemia. Statins or PCSK9 inhibitors for primary prevention of ASCVD are acceptable.

   * Fibrates (e.g., fenofibrate, clofibrate, gemfibrozil)
   * High-dose niacin (>100 mg daily)
7. Known, documented history, at the time of screening, of any of the following medical conditions:

   i. Pancreatic pathology ii. Significant cardiovascular diseases (N.B. uncomplicated hypertension is not exclusionary) iii. Chronic kidney disease, Stage 3 or higher (estimated glomerular filtration rate < 60 mL / min / 1.73 m2), of any cause iv. Advanced or severe liver disease v. Gallstone disease vi. Chronic viral illness including human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) (N.B. diagnosis based only on medical history; we will not test for any of these viruses at any point in this study) vii. Active malabsorptive conditions viii. Active seizure disorder (including controlled with antiepileptic drugs) ix. Psychiatric diseases causing functional impairment that have been decompensated within 1 year or require use of drugs associated with significant weight gain/metabolic dysfunction x. Other endocrinopathies (e.g., Cushing syndrome, adrenal insufficiency) xi. Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation xii. Bleeding disorders, including due to anticoagulation, or significant anemia (see above) xiii. Dysautonomia, including post-vagotomy xiv. Active malignancy, or hormonally active benign neoplasm, except for non-melanoma skin cancer or differentiated thyroid cancer (AJCC Stage I only)
8. Clinical concern for increased risk of volume overload, including due to medications and/or heart/liver/kidney problems, as listed above
9. Clinical concern for increased risk of hypokalemia, including low potassium on screening labs (i.e., below lower limit of normal), use of certain medications, or any medical conditions listed above
10. Use of certain medications currently or within 90 d prior to screening:

    i. Prescribed medications used for any of the indications in the preceding list of excluded conditions, or their use within 90 d prior to screening, except allowances for:

    • Use of drugs prescribed for indications other than the exclusionary diagnoses/purposes listed above (e.g., antiepileptic drugs used for non-seizure indications, angiotensin converting enzyme inhibitor (ACEi)/angiotensin receptor blocker (ARB) used for uncomplicated hypertension rather than for congestive heart failure, etc.)

    •• Note, as above, that antidiabetic drugs except metformin for any indication within 90 d of screening are excluded ii. Oral or parenteral corticosteroids (at greater than prednisone 5 mg daily, or equivalent) for more than 3 days within the previous 90 days; topical and inhaled formulations are permitted iii. Fludrocortisone iv. Opioids other than dextromethorphan for cough
11. History of certain weight-loss (bariatric) surgery, including:

    i. Roux-en-Y gastric bypass ii. Biliopancreatic diversion iii. Restrictive procedures (lap band, sleeve gastrectomy) performed within the past 6 months
12. Clinical concern for alcohol overuse, including recent documented history or phosphatidylethanol ≥ 0.05 µmol/L at screening and/or participant report of regularly consuming more than 2 drinks per day for males or 1 drink per day for females.
13. Positive urine drug screen, with exceptions for:

    i. Lawfully prescribed medications ii. Marijuana/THC positivity, provided that the participant agrees not to use it during the same period that they will abstain from alcohol
14. History of severe infection or ongoing febrile illness within 30 days of screening
15. Any other disease, condition, or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
16. Known allergy/hypersensitivity to any component of the medicinal product formulations (including soy or dairy), IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
17. Concurrent enrollment in another clinical study of any investigational drug therapy within 6 months prior to screening or within 5 half-lives of an investigational agent, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Plasma glucose (absolute values) (units: mg/dL) | Up to 425 minutes from the start of the procedure.
  Goal is first to clamp insulin infusion rate to maintain mean basal fasting plasma glucose during the basal titration phase, and then during the intervention phase to observe the glucose levels that result from altering the basal IIR.
Plasma glucose (relative/change) (units: fold difference and/or ∆mg/dL relative to previous time points) | Up to 425 minutes from the start of the procedure.
  Goal is first to clamp insulin infusion rate to maintain mean basal fasting plasma glucose during the basal titration phase, and then during the intervention phase to observe the impact of altering the basal IIR on glycemia.
Serum insulin (absolute values) (units: micro-international units per milliliter (µIU/mL)) | Up to 425 minutes from the start of the procedure.
  Investigators will assess the insulin levels attained at the basal IIR, and at each stepwise reduction in IIR during the intervention phase.
Serum insulin (relative/change) (units: fold difference and/or ∆ µIU/mL relative to previous time points) | Up to 425 minutes from the start of the procedure.
  Investigators will compare the baseline insulin level to that attained at the basal IIR, as well as comparing to the change in insulin level that occurs with alterations in the IIR during the intervention phase.
Serum C-peptide (absolute values) (units: ng/mL) | Up to 425 minutes from the start of the procedure
  Suppression of endogenous insulin by octreotide during pancreatic clamp is expected to result in a fall in C-peptide levels to near zero.
Serum C-peptide (relative/change) (units: fold difference and/or ∆ µIU/mL relative to previous time points) | Up to 425 minutes from the start of the procedure
  Suppression of endogenous insulin by octreotide during pancreatic clamp is expected to result in a fall in C-peptide levels to near zero.

SECONDARY OUTCOMES:
Serum or plasma triglyceride (TG) (absolute values) (units: mg/dL) | Up to 425 minutes from the start of the procedure
  TG levels in serum reflect hepatic synthesis/storage and very low-density lipoprotein (VLDL) secretion.
Serum or plasma triglyceride (TG) (relative/change) (units: fold difference and/or ∆mg/dL relative to previous time points) | Up to 425 minutes from the start of the procedure
  TG levels in serum reflect hepatic synthesis/storage and VLDL secretion.
Serum or plasma free fatty acid (FFA) (absolute values) (units: mg/dL) | Up to 425 minutes from the start of the procedure
  FFA levels reflect adipose tissue lipolysis and its response to insulin and counterregulatory hormones.
Serum or plasma free fatty acid (FFA) (relative/change) (units: fold difference and/or ∆mg/dL relative to previous time points) | Up to 425 minutes from the start of the procedure
  FFA levels reflect adipose tissue lipolysis and its response to insulin and counterregulatory hormones.
Serum or plasma apolipoprotein B (ApoB) (absolute values) (units: mg/dL) | Up to 425 minutes from the start of the procedure
  ApoB level is a surrogate for triglyceride-rich lipoproteins, especially hepatic VLDL.
Serum or plasma apolipoprotein B (ApoB) (relative/change) (units: fold difference and/or ∆mg/dL relative to previous time points) | Up to 425 minutes from the start of the procedure
  ApoB level is a surrogate for triglyceride-rich lipoproteins, especially hepatic VLDL.
Plasma glucose kinetics: rate of appearance (units: mg/kg/min) | Measured every 5 minutes x 4 at the end of each steady-state IIR period, up to 425 minutes from the start of the procedure
  Calculated from D2G tracer enrichment by the Steele equations.
Plasma glucose kinetics: rate of disappearance (units: mg/kg/min) | Measured every 5 minutes x 4 at the end of each steady-state IIR period, up to 425 minutes from the start of the procedure
  Calculated from D2G tracer enrichment by the Steele equations
Plasma glucose kinetics: endogenous glucose production (units: mg/kg/min) | Measured every 5 minutes x 4 at the end of each steady-state IIR period, up to 425 minutes from the start of the procedure
  Calculated from D2G tracer enrichment by the Steele equations

OTHER OUTCOMES:
Serum/plasma glucagon (absolute values) (units: ng/L) | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous glucagon replacement.
Serum or plasma glucagon (relative/change) (units: fold difference and/or ∆ng/L relative to previous time points) | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous glucagon replacement.
Serum or plasma growth hormone (absolute values) (units: ng/mL) | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous rhGH replacement.
Serum or plasma growth hormone (relative/change) (units: fold difference and/or ∆ng/mL relative to previous time points) | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous rhGH replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R. Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Blood samples will be banked in our Insulin Resistance Biobank and will be made available to other researchers for legitimate research purposes upon request. Associated data will be shared along with specimens in the smallest possible quantity and on a need-to-know basis. No Protected Health Information (PHI) will ever be disclosed to other researchers. All requests will be reviewed by the PI for scientific merit and samples/data will be transferred only upon completion of an Institutional Review Board-approved Material Transfer Agreement (MTA) and/or Data Use Agreement (DUA), as appropriate.
Supporting Information: Study Protocol
Time Frame: Indefinitely following study completion.
Access Criteria: All requests will be reviewed by the PI for scientific merit and samples/data will be transferred only upon completion of a MTA or DUA, as appropriate. No PHI will be disclosed or shared.